CLINICAL TRIAL: NCT01683968
Title: Diastolic Dysfunction in Sickle Cell Disease During Vaso-occlusive Crisis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: King Abdullah International Medical Research Center (Other)
Collaborators: King Abdulaziz Medical City (Other Government)
Responsible Party: Principal Investigator, Abdulsalam Alaithan, CONSULTANT INTENSIVEST AND PULMONOLOGIST, King Abdulaziz Medical City
Other Study IDs: RE11/027
Record Dates: First submitted 2012-09-08; First posted 2012-09-12 (Estimated); Last update posted 2012-09-13 (Estimated); Status verified 2012-09

CONDITIONS: Sickle Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Sickle cell: Patient who are admitted with sickle cell crises

SUMMARY:
This study is designed to investigate the presence and absence of abnormal heart muscle contractions during sickle cell crises.

You will be asked to do echocardiography during and after your admission to the hospital. We will compare tow pictures and study the differences.

DETAILED DESCRIPTION:
Sickle cell disease (SCD) is a common genetic disorder of hemoglobin synthesis. Although sickle disease is globally spread it is more common in sub-Saharan Africa, India, Saudi Arabia and Mediterranean countries1. In Saudi Arabia, the prevalence of sickle cell disease id 24 per 10,000 with a higher prevalence in eastern province 145 per 10,0002.

The vaso-occlusive crisis is the principal presentation of SCD3. Acute pain is the primary and most common symptom of vaso-occlusive crisis4. Pain management and fluid resuscitation are the mainstay therapy for the treatment of vaso-occlusive crisis5. Pulmonary edema has been reported as a complication of fluid therapy during acute crisis management6. However, the exact mechanism of pulmonary edema in this population is not fully understood. Recent studies have demonstrated the presence of diastolic dysfunction in patients with SCD. Diastolic dysfunction was reported in 18% of patients with SCD7. These studies were performed when the patients were not in vaso-occlusive crisis.

Objectives of the Study:

Study hypothesis: Previous studies have shown that the prevalence of diastolic dysfunction is 18% (14-17). These studies have evaluated the general population of SCD without the distention whether these evaluations were made during the acute crisis or not. Others have also demonstrated increased pulmonary pressure in this patient population (32,33) . We hypothesize that the degree of diastolic dysfunction gets worse during acute vaso-occlusive crisis and may translate to higher pulmonary artery pressure and/or development of pulmonary edema during fluid therapy Study Area/Setting King Abdulaziz Hospital Alhasa

The primary objective if the study is to evaluate the presence and the degree of diastolic dysfunction during the Vaso-occlusive crisis of sickle cell disease. This will be achieved by evaluating multiple echocardiography parameters in accordance with the American Society of Echocardiography (ASE) Guidelines 10. These parameters include: Mitral valve inflow Hemodynamic E/A ratio and deceleration time(DT), septal and lateral mitral annular velocities (e')by tissue Doppler, and left atrial volume. According to these parameters the diastolic function can be evaluated as normal or abnormal. If abnormal then the diastolic dysfunction can be subsequently classified into impaired relaxation, pseudo-normalization and restrictive physiology(10-13). These parameters are age related (see table 1). The La volume will be measured by area by Biplane area-length method according to the formula (0.85) *( A1*A2/L) Where is A1 is left atrial volume in 4chamer view, A2 is left atrial volume in 2 chamber view and L is the length measured form the back wall of the left atrium to the mitral valve hinge point(14).

The grading of diastolic dysfunction will be as follows:

1. Grade I (impaired relaxation): E/A< 0.8, DT>200 ms, E/e' </= 8 and LA volume >34 ml/m2.
2. Grade II (pseudo-normalization): E/A=0.8- 1.5, DT= 160-200 ms, E/e' = 9-12 and LA volume >34 ml/m2.
3. Grade II (restrictive physiology): E/A >2, DT<160 ms, E/e'>/=13 and LA volume >34 ml/m2.
4. In case of overlap of these parameters so that no single category can be assigned the diastolic function will be categorized as abnormal.

The pulmonary artery pressure will be determined non-invasively on echocardiography by measuring tricuspid regurgitation jet velocity and adding the estimated right atrial pressure (15-17).

Pulmonary edema will be diagnosed either clinically by the presence of fine inspiratory crepitations on chest examination and high jugular venous pressure, and radio graphically by the presence of venous congestion and/or Kerley B-lines after confirming the finding by consultant radiologist oncall (18-20).

The vaso-occlusive crisis will be diagnosed clinically be the presence of the classical symptoms of pain and dehydration in the absence of alternative diagnosis (21-23).

Controls: The follow up echo (second echo) will be used as a baseline to compare the findings in the acute crisis to. As it is difficult to decide who of the patients with SCD will develop the acute crisis, we decided to recruit patients presenting in acute crisis and redo the echo as a follow up and use the follow up echo as a baseline looking at the same parameters.

Study Design Prospective cross sectional study Sample Size 50% probability of having the outcome of interest. Assuming 10% drop rate the number of needed subject would be 216 patients to achieving 95% confidence, 7 % margin of error.

Sampling Technique A consecutive inpatient admission to medical ward will be enrolled in the study according to inclusion and exclusion criteria mentioned above.

Data Management and Analysis Plan The SPSS for Windows 19.0 programme (SPSS Inc, Chicago, Illinois) will be used for statistical analysis. The chi-square test was used to analyze categorical variables and the Student's t test was used to analyze parametric variables. A p-value of 0.05 or less was considered statistically significant.

ELIGIBILITY:
Inclusion criteria:

1. Patients older than 18 years
2. Diagnosis of acute vaso-occlusive crisis due to sickle cell disease.
3. Informed consent

Exclusion criteria:

1. Congenital heart disease
2. Long standing hypertension

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patient admitted to the hospital with vaso-occlusive crisis
Sampling Method: Non-Probability Sample
Enrollment: 216 (Estimated)
Dates: Start 2012-09; Primary Completion 2015-10 (Estimated); Study Completion 2015-10 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- King Abdulaziz Hospital, Al-Ahsa, EP, Saudi Arabia